CLINICAL TRIAL: NCT07060053
Title: The Effect of Oil Pulling on Oral Health-related Quality of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Christine Zürcher (Other)
Responsible Party: Sponsor-Investigator, Christine Zürcher, Dr., Medical University Innsbruck
Organization: Medical University Innsbruck (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: EK Nr 1117/2022
Record Dates: First submitted 2025-05-19; First posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-05

CONDITIONS: Oral Health Related Quality of Life
MeSH Terms: interventions — Sesame Oil

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- sesame oil (Experimental): 8 weeks oil pulling with 15 ml of sesame-based oil for 15min every morning
  Interventions: Other: sesame oil
- distilled water (Other): 8 weeks rinsing with 15ml of distilled water for 15min every morning
  Interventions: Other: distilled water

INTERVENTIONS:
Other: sesame oil — 15min of oil pulling with 15ml sesame-based oil for 8 weeks
  Arms: sesame oil
Other: distilled water — 15min rinsing with 15ml distilled water for 8 weeks
  Arms: distilled water

SUMMARY:
To date, there are no studies assessing the impact of mouth rinses on the oral health-related quality of life in healthy patients with gingivitis. Thus, this study aimed to assess the effect of oil pulling on the OHRQoL using the 14-item OHIP questionnaire (OHIP-14). The null hypothesis stated, that there would be no significant difference in OHIP-14 scores between individuals with gingivitis performing oil pulling with sesam-based oil and those using distilled water over an eight-week period.

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years
* contractual capability
* the presence of ≥ 10 teeth,
* community periodontal index of treatment needs (CPITN) grade 1 or 2

Exclusion Criteria:

* missing consent
* community periodontal index of treatment needs (CPITN) grade 0, 3 or 4
* pregnancy or breastfeeding
* systemic diseases or conditions that are associated with an increased risk of infection or necessitate concomitant antibiotic therapy with dental treatment
* mental and behavioral disorders that impede (verbal) communication
* allergy against sesame(oil)
* intake of antibiotics 6 months prior to or during study duration
* intake of medication potentially influencing gingival inflammation or bleeding (e.g. anticoagulants, cortisone)
* infectious diseases (e.g. HIV, hepatitis B or C)
* fixed orthodontic appliances
* ongoing oil pulling or mouth rinsing
* adult guardianship
* insufficient nasal breathing

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-05-04 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

PRIMARY OUTCOMES:
OHIP | first follow up after 4 weeks, full study duration 8 weeks
  The Oral Health Impact Profile-14 (OHIP-14), a questionnaire with 14 questions, evaluates the impact of oral health on quality of life across seven domains: functional limitation, physical pain, psychological discomfort, physical disability, psychological disability, social disability, and speech limitation. Each of the 14 items is rated on a 5-point Likert scale, ranging from 0 (never) to 4 (very often). A total score of zero reflects the best possible oral health-related quality of life, while a score of 56 indicates the poorest. The validated German version of the questionnaire was used

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University Innsbruck, Innsbruck, Tyrol, Austria

IPD SHARING:
Plan to Share IPD: No